CLINICAL TRIAL: NCT07185841
Title: A Multicenter, Open-label, Phase I/II Study to Evaluate the Safety, Pharmacokinetics and Efficacy of Oral HX9428 Tablets in Subjects With Wet Age-related Macular Degeneration (wAMD)
Brief Title: Safety and Efficacy of Oral HX9428 Tablets in Subjects With Wet Age-related Macular Degeneration (wAMD)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fujian Haixi Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HXP056-CTPI-01
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Wet Age-related Macular Degeneration (AMD)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HX9428 tablet (Experimental): Escalating dose of HX9428 tablet starting at 5mg once a day.
  Interventions: Drug: HX9428 tablet

INTERVENTIONS:
Drug: HX9428 tablet — Subjects will receive HX9428 orally every day. The total treatment period is tentatively set at 25 weeks..

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of Oral HX9428 tablets in patients with wet age-related macular degeneration(wAMD)

DETAILED DESCRIPTION:
This is a Multicenter, Open-label, Phase I/II Study to Evaluate the Safety, Pharmacokinetics and Efficacy of Oral HX9428 tablets in Subjects with Wet Age-related Macular Degeneration (wAMD). The study consists of 2 segments: Phase I and Phase II. Phase I will evaluate the safety and tolerability of HX9428 administered as single and multiple oral doses; dose escalation will follow a 3 + 3 design with overdose control. If evidence of efficacy is observed at any dose level during Phase I, a parallel Phase II study may be initiated while dose-escalation in Phase I continues. In Phase II, the daily dose of HX9428 will not exceed the Maximum Tolerated Dose (MTD) established in Phase I; dosing frequency will be once daily (QD) or every other day (QOD).The primary objective of Phase II is to assess the preliminary efficacy of HX9428 tablets under these regimens.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria for study entry:

  1. Age ≥50 years and ≤80 years (Phase I), Age ≥50 years and ≤85 years (Phase II) at the time of signing informed consent, male or female;
  2. Active choroidal neovascularization (CNV) secondary to AMD, as evidenced on fluorescein fundus angiography (FFA) and optical coherence tomography (OCT) (Active CNV is defined as the presence of subretinal or intraretinal fluid or leakage); A total lesion size of <12 disc areas on FFA ;
  3. Treatment-naive , or previous anti-VEGF treatment that was effective and discontinued for more than 3 months, with OCT evidence of subretinal fluid or cystoid macular edema;
  4. ETDRS BCVA 19 to 78 letters in the study eyes( corresponding to a Snellen equivalent of approximately 20/32 to 20/400) ;
  5. Other protocol-specified inclusion criteria may apply

Exclusion Criteria:

* Subjects who meet any of the following criteria will be excluded from this study:

  1. Subjects diagnosed with polypoidal choroidal vasculopathy by Indocyanine Green(ICG) angiography who are at high risk of massive hemorrhage;
  2. On FFA/CFP: subretinal hemorrhage of >50 % of the total lesion area or that involves the fovea; fibrosis or atrophy of >50 % of the total lesion area or that involves the fovea;
  3. CNV due to causes other than AMD;
  4. Any condition in the study eye that could compromise best-corrected visual acuity;
  5. Active ocular inflammation or infection in either eye or a history of idiopathic or autoimmune-related uveitis;
  6. Refractive error exceeding -6.00 D spherical equivalent;
  7. Ocular surgery performed in the study eye within 90 days before screening;
  8. Previous treatment with photodynamic therapy (within 120 days of screening), external-beam radiotherapy, macular laser photocoagulation, macular surgery, or transpupillary thermotherapy;
  9. Systemic anti-VEGF therapy administered within 90 days before the first dose;
  10. Pregnant or lactating women;
  11. Known hypersensitivity or contraindication to any study-related procedure drugs;
  12. History of severe cardiac disease, symptomatic congestive heart failure, unstable angina, acute coronary syndrome, myocardial infarction, coronary revascularization, thrombotic event, or bleeding episode within 6 months prior to the start of study drug, uncontrolled hypertension (systolic blood pressure> 150 mmHg and/or diastolic blood pressure > 100 mmHg on optimal medical therapy), or ventricular arrhythmia requiring ongoing treatment;
  13. Stroke within 12 months or transient ischemic attack within 6 months of enrolment；
  14. Poorly controlled diabetes (HbA1c ≥ 12 %);
  15. Other protocol-specified exclusion criteria may apply.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-01-07 (Estimated)

PRIMARY OUTCOMES:
Phase I : Dose-Limiting Toxicity (DLT) | Week 4
  Dose-limiting toxicity (DLT) refers to a drug-related toxicity during treatment with the drug, the severity of which is clinically unacceptable, limiting the further escalation of drug dose
Phase II： Mean change of letters from baseline in Best Corrected Visual Acuity(BCVA) | week 25
  Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity.

SECONDARY OUTCOMES:
Mean change from baseline in Central Subfield Thickness（CST） | week 25
  Evaluated by Optical Coherence Tomography (OCT). The higher values means worse outcome.
Proportion of patients gaining at least 15/10/5 letters from baseline in the BCVA | Week 25
  Best Corrected Visual Acuity (BCVA) was measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity.
Mean change from baseline in the total area of CNV and the total area of fluorescein leakage | Week 25
  Evaluated by Fundus Fluorescein Angiography (FFA)
Pharmacokinetic (PK) profile | Week 4
  Study the change of HX9428 drug concentration in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Hong Dai, Principal Investigator — Beijing Hospital
Locations (1):
- Beijing Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No